CLINICAL TRIAL: NCT04037956
Title: A Perspective Study to Compare the Tubeless NOSES and Traditional Laparoscopic Radical Resection in Rectosigmoid Cancers (CORNER)
Brief Title: Tubeless NOSES Versus Laparoscopic Radical Resection for Rectosigmoid Cancers
Acronym: CORNER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanxin Luo,MD, Deputy Chief Physician, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SixthSunYetSen-Lyx
Record Dates: First submitted 2019-07-16; First posted 2019-07-30 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Tubeless NOSES; Traditional Laparoscopic Radical Resection; Rectosigmoid Cancers
Keywords: Tubeless NOSES; traditional laparoscopic radical resection; Rectosigmoid Cancers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tubeless NOSES (Experimental): Patients receive Tubeless NOSES.
  Interventions: Procedure: Tubeless NOSES
- traditional laparoscopic (Active Comparator): Patients receive traditional laparoscopic radical resection.
  Interventions: Procedure: traditional laparoscopic radical resection

INTERVENTIONS:
Procedure: Tubeless NOSES — The whole procedures undergo by total laparoscopic surgery with no specimen extraction incision in the abdominal wall. The specimen then will be removed through natural orifice such (anal).
  Arms: Tubeless NOSES
Procedure: traditional laparoscopic radical resection — The traditional laparoscopic operation undergo and then a small incision(5-8cm) is made in the middle of the lower abdominal wall to remove the specimen.
  Arms: traditional laparoscopic

SUMMARY:
This study is designed to evaluate the short-term and long-term results after Tubeless NOSES for the resection of Rectosigmoid Cancers compared with traditional laparoscopic radical resection.

DETAILED DESCRIPTION:
This is a randomized, single-center, open-label, non- inferiority study designed to evaluate the safety, efficacy and potential benefits of Tubeless NOSES compared with traditional laparoscopic radical resection in approximately 458 subjects with Rectosigmoid Cancers.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed Rectosigmoid Cancers
2. Clinical stage at T 1-3 N0-2 M0
3. Tumors on peritoneal reflection，Tumor size is no more than 3 cm
4. Eastern Cooperative Oncology Group (ECOG) scale is 0-2
5. American Society of Anesthesiologists (ASA) score is Ⅰ-Ⅲ
6. BMI ≤ 30 kg/m2
7. Subjects must be willing and able to comply with scheduled visits, treatment schedule,and laboratory testing.

Exclusion Criteria:

1. Heart, lung, liver or renal or any organ function that are intolerance for surgery
2. History of treated colorectal malignant disease
3. Subjects with medical condition, such as intestinal obstruction, intestinal perforation, bleeding, requires emergency surgery
4. Subjects with previous malignancies
5. History of inflammatory bowl disease(IBD) or familial adenomatous polyposis (FAP)
6. Treatment with any other clinical trial within 28 days prior to randomization
7. History of severe mentally disease
8. pregnant or lactating women
9. The researchers believe that the patients are unsuitable to participate in the researchers with other cases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival rate | 36 months after surgery

SECONDARY OUTCOMES:
5-year overall survival rate | 60 months after surgery
Incidence of postoperative complications | 1 month after surgery
  All postoperative complications in the perioperative period will be classified by the Clavien-Dindo classification.
the functional outcome of defecation | 60 months after surgery
  Anal incontinence was evaluated using the Wexner Continence Grading Scale , the score being calculated after the patients' completion of a daily defecatory questionnaire. Range is from 0 (normal continence) to 20 (maximum incontinence with maximum disturbance of lifestyle).
the operation time | in the perioperative period
  The descriptive unit would be minute (min).
the blood loss during the operation | in the perioperative period
  The descriptive unit would be millilitre (ml)
Postoperative recovery of intestinal peristalsis | in the perioperative period
  The descriptive unit would be hour (h).
Pain score | in the perioperative period
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured.It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms.For example, the amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain ( from 0 to 10).
number of cases converted to laparotomy | in the perioperative period
  The procedure for cases who underwent traditional laparoscopic radical resection for those who cannot be done with traditional laparoscopic radical resection or Tubless NOSES and convert to laparotomy as a result，these should be recorded and compared within two experimental arms.
the mean postoperative hospitalization day | in the perioperative period
  The descriptive unit would be day (d).

CONTACTS AND LOCATIONS:
Overall Officials: Yanxin Luo, phD, Study Chair — The Sixth Affiliate Hospital of Sun Yat-Sen University
Locations (1):
- The Sixth Affiliate Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.